CLINICAL TRIAL: NCT01532895
Title: Clinical Usefulness and Quality of Life of OROS Hydromorphone in Strong Opioid-Naïve Cancer Pain Patients; Multicenter, Prospective, Open-Label and Observational Study
Brief Title: Clinical Usefulness and Quality of Life of OROS Hydromorphone in Patients Who Have Not Been Treated With a Strong Opioid
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100741; 42801PAI4013 (Other: Janssen Korea, Ltd., Korea); HYD-KOR-5011 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Pain
Keywords: Pain; Cancer pain; Hydromorphone; Hydromorphone OROS; Narcotic analgesics; Opioid-naive
MeSH Terms: conditions — Pain; Cancer Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hydromorphone HCI OROS
  Interventions: Drug: Hydromorphone HCI OROS

INTERVENTIONS:
Drug: Hydromorphone HCI OROS — type= exact number, unit= mg, number=4, form= tablet, route= oral use. One tablet administered once a day. The dose may be increased if the level of pain increases or if the pain-killing effect is insufficient.

SUMMARY:
The primary purpose of this study is to evaluate the usefulness of hydromorphone to treat cancer pain in patients who have not been treated with a strong opioid.

DETAILED DESCRIPTION:
This is a multicenter, prospective, open-label (all people know the identity of the intervention) and observational study. Patients selected for the proposed study are patients complaining of cancer pain who visit or are hospitalized at the research centers during the study, who are not being treated with strong continuous opioid (narcotic medication used against the pain), and who require cancer pain control with hydromorphone, at the investigator's discretion. The study will evaluate the changes in pain relief, level of sleep deprivation, and the patients' quality of life before and after administration of hydromorphone.

ELIGIBILITY:
Inclusion Criteria: - Patients who complain of cancer pain and who require administration of hydromorphone HCl - Patients who can follow the requirements of the overall study, including completion of filling out the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, at the investigator's discretion - Signed informed consent Exclusion Criteria: - Patients who received strong continuous narcotic analgesics (eg morphine, fentanyl, oxycodone, hydromorphone) within 4 weeks prior to administration of the study drug - Patients who have a medical history of receiving drugs in the past or currently, or of drug abuse - Patients who did not agree to conduct the approved methods for contraception during the study - Patients who have sustained injuries in physical functions or diseases which may cause abnormalities in absorbing the study drug, excessive accumulation and metabolic or elimination disorder - Patients who are receiving Monoamine Oxidase Inhibitors (MAO) inhibitors or who are within 2 weeks from discontinuation - Patients who need to be excluded based on precautions in the user manual of the study drug, notice and contradictions, at the investigator's discretion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean cancer patients having cancer pain who visit or are hospitalized at the research centers during the study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The ratio of patients with % PID (Pain Intensity Difference) over 30% of patients from the first evaluation date until the third evaluation date, following the administration of hydromorphone HCI to cancer pain patients | Baseline and at approximately Day 57

SECONDARY OUTCOMES:
Changes in the Karnofsky Performance Rating Scale (KPRS) | Baseline, and at approximately Days 29 and 57
  The KPRS measures the physical functions of cancer patients, and indicates the feasibility of daily life by 10% units from 0% (death) to 100% (normal status in which patients can do activities to the level before disease without limitations).
Change in pain relief (%) | Baseline, and at approximately Days 29 and 57
  How much pain was relieved by the pain therapy or medication for the last 24 hours, using %: 0%= nothing reduced and 100%= completely reduced.
Frequency of awakening | Baseline, and at approximately Days 29 and 57
  Check whether patients experienced awakening during sleep caused by pain for the last 1 week or not, and measure the frequency (1 = once, 2 = twice, 3 = 3 times, 4 = more than 4 times, 5 = not woken, 6 = never slept).
Level of sleep inconvenience | Baseline, and at approximately Days 29 and 57
  Measure the level of sleep inconvenience that patients experienced due to pain for the last 1 week using the Numeric Rating Scale (NRS); 0 = not causing inconvenience, 10 = completely causing inconvenience.
Satisfaction with sleep | Baseline, and at approximately Days 29 and 57
  Indicate the overall satisfaction with sleep by improving sleep disturbance caused by pain for the last 1 week using the Numeric Rating Scale (0 "never satisfied" on the left end; 10 "very satisfied" on the right end).
Quality of life assessment measured by the EORTC QLQ-C15 PAL | Baseline, and at approximately Days 29 and 57
  The EORTC (European Organization for Research and Treatment of Cancer) QLQ-C15 (Quality of Life Questionnaire Core 15) is a commonly used questionnaire to assess the quality of life of cancer patients taking paliative medicine. This questionnaire consists of questions measuring physical, role, emotional, cognitive and social functions, and answers are given based on a 4-point scale, from 1 (not at all) to 4 (very much so).
Investigator's Global Assessment | At approximately Days 29 and 57
  The investigator's global assessment is used to assess how effective the study drug was for the patients after administration of the study drug since the last evaluation date. It is measured by the investigator from the investigator's point of view as 1 = not effective, 2 = normal l, 3 = effective, 4 very effective, and 5 = extremely effective.
Patient's Global Assessment | At approximately Days 29 and 57
  The patient's global assessment is used to assess how effective the study drug was for the patients after administration of the study drug since the last evaluation date. It is measured by the patient from the patient's point of view as 1 = not effective, 2 = normal, 3 = effective, 4 = very effective, and 5 = extremely effective.
CGI-I (Clinical Global Impression - Improvement) | At approximately Days 29 and 57
  Evaluate how much patients have improved compared with the conditions of patients at baseline, from 1 (very much improved) to 7 (greatly deteriorated).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (11):
- South Korea (11):
  - Ansan
  - Busan
  - Cheongju-si
  - Daegu
  - Hwasun Gun
  - Incheon
  - Pusan
  - Seognam-Si, Kyungki-Do
  - Seoul
  - Suwon
  - Wonju-Shi